CLINICAL TRIAL: NCT05339048
Title: Observational Study for the Analysis of Associations Between Cardiovascular and Respiratory Diseases in a Cohort of Latin American Adults
Brief Title: The Cartagena Cohort Study
Acronym: CaReS
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidad de Cartagena (Other)
Collaborators: The Administrative Department of Science, Technology and Innovation, Colciencias (Other); National Center for Research in Chronic Diseases, Colombia (Unknown); Johns Hopkins Bloomberg School of Public Health (Other); Universidad Catolica de Cordoba (Unknown); University of Chile (Other); Universidad de Sucre (Unknown); Universidad del Magdalena (Other)
Responsible Party: Principal Investigator, Gustavo Mora Garcia, Associate professor, Universidad de Cartagena
Other Study IDs: CCS
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases; COPD; Lung Function Decreased; Atherosclerosis
Keywords: Low and middle income countries; Non-communicable diseases; Latin America; Cardio-respiratory disease
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Atherosclerosis; Noncommunicable Diseases | interventions — Diet; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole human DNA from blood samples. Microbiome DNA sample from oral-pharyngeal mucose samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General group: 18-80 years old adults from the Colombian Caribbean Coast.
  Interventions: Genetic: Genetic risk variants; Other: Diet; Behavioral: Physical activity; Other: Socio-economic conditions

INTERVENTIONS:
Genetic: Genetic risk variants — Exposure: Genetic predisposition to complex diseases.
Other: Diet — Exposure: dietary intake of unhealthy foods known to be associated with higher prevalence of respiratory and cardiovascular diseases.
Behavioral: Physical activity — Exposure: frequency of moderated or intense physical activity, and daily exposure to sedentary behavior.
Other: Socio-economic conditions — Exposure: socio-economic vulnerability indexes associated with higher prevalence of respiratory and cardiovascular diseases (including household conditions, accessibility to health care services, among others).

SUMMARY:
Cardiovascular and respiratory diseases are the first and third cause of death, respectively. Cardiovascular risk is known to increase in groups with impaired lung function; however, the mechanisms behind this association are not fully understood. The aim of CaReS is to elucidate the shared pathophysiology of impaired lung function and cardiovascular risk, and to investigate the risk factors associated with them.

The CaReS Cohort Study includes adults (18-80 years old) from Cartagena de Indias, a tropical city on Colombian Caribbean Coast, where recent population admixture settled a three-hybrid genetic structure (European, African and Ameridian ancestry). At baseline, the cohort will generate extensive data on -omics (e.g., genomics, transcriptomics, metabolomics, and epigenomics), socio-economic wellbeing, lifestyle, medical history, cardiometabolic, inflammatory and liver function markers, as well as objective measures of ventilatory and cardiovascular performance.

The cohort will collect data every three years, for a total period of ten years. Prospective risk of cardiovascular disease and chronic obstructive pulmonary disease (COPD) will be investigated, and their risk factors. Throughout the study period, changes in prevalence, and interactions of various risk factors with these changes will also be ascertained.

A predictive risk score for cardiovascular and chronic respiratory disability will be built, using cross-sectional and longitudinal data.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Native from Colombian Caribbean Coast

Exclusion Criteria:

* Pregnant women
* Walking physical disability
* Cognitive disability
* Patients under treatment for any type of cancer
* Clinical record of primary chronic endocrine disease
* Clinical record of major respiratory tract surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults, men and women, living on Colombian Caribbean Coast.
Sampling Method: Non-Probability Sample
Enrollment: 619 (Estimated)
Dates: Start 2020-10-03 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2034-10-02 (Estimated)

PRIMARY OUTCOMES:
Atherosclerosis | baseline - 10 years (end of follow up)
  Carotid atheroma identified by eco-doppler imaging test
Acute cardiovascular event | 2nd year (first follow up) - 10 years (end of follow up)
  Record of acute coronary heart disease, miocardipathy, and ischemic or hemorragic cerebrovascular event.
Chronic airflow obstruction | baseline - 10 years (end of follow up)
  Obstruction patterns in post-bronchodilator spirometry.
Metabolic syndrome | baseline - 10 years (end of follow up)
  Pathologic findings for blood pressure, triglycerides, HDLc, serum glucose, and/or enlarged waist circumference (three or more of this criteria found simultaneously)

SECONDARY OUTCOMES:
Chronic Obstructive Pulmonary Disease (COPD) | baseline - 10 years (end of follow up)
  Diagnosis of by lung function test (post-bronchodilator spirometry) and/or clinical criteria
Hypertension | baseline - 10 years (end of follow up)
  Primary high blood pressure according to clinical criteria
Type 2 Diabetes Mellitus | baseline - 10 years (end of follow up)
  Abnormal results in fasting serum glucose test and/or HbA1c test.
Dyslipidemia | baseline - 10 years (end of follow up)
  High serum cholesterol, triglycerides or LDLc; and/or low HDLc

CONTACTS AND LOCATIONS:
Overall Officials: GUSTAVO J MORA-GARCIA, PhD, Principal Investigator — Universidad de Cartagena; VANESSA GARCIA-LARSEN, PhD, Study Director — BLOOMBERG SCHOOL OF PUBLIC HEALTH JOHNS HOPKINS UNIVERSITY; MARIA S RUIZ-DIAZ, PhD, Study Chair — NATIONAL CENTER FOR RESEARCH IN CHRONIC DISEASES
Locations (1):
- Universidad de Cartagena, Cartagena, Departamento de Bolívar, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Documents (i.e., study protocol, informed consent, and laboratory test) and study database are being save on a secure server at https://redcap.unicartagena.edu.co/redcap/
  Sharing of study protocol, statistical analysis plan and analytic code is awaiting to be discussed by the research team.